CLINICAL TRIAL: NCT01610882
Title: Panda: Evaluation of a Smartphone-based Perioperative Pain Assessment Tool
Acronym: Panda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Mark Ansermino, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: H12-01273
Record Dates: First submitted 2012-05-29; First posted 2012-06-04 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Acute Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Panda first (Other): Panda evaluation of post-operative pain first, followed by manual method of pain assessment.
  Interventions: Device: Panda first followed by manual pain assessment
- Manual first (Other): Manual evaluation of post-operative pain first followed by Panda pain assessment.
  Interventions: Device: Manual first followed by Panda pain assessment

INTERVENTIONS:
Device: Panda first followed by manual pain assessment — Panda is a smart-phone based application designed to assess post-operative pain; manual method involves use of CAS/FPS-R on paper. Panda will be used first, manual method 5 mins later.
  Arms: Panda first
Device: Manual first followed by Panda pain assessment — Panda is a smart-phone based application designed to assess post-operative pain; manual method involves use of CAS/FPS-R on paper. Manual method will be used first, Panda 5 mins later.
  Arms: Manual first

SUMMARY:
This study will evaluate Panda, a smartphone-based pain assessment tool. During a child's recovery from surgery, a Post-Anesthetic Care Unit nurse will assess their pain, which helps determine what medication they need. Traditionally, this involves asking the child to rate their pain on a scale from 1 to 10, by moving a slider along a coloured scale or pointing to one of a series of faces on a piece of card. The Panda uses the same methods, but presents them on a smartphone screen. Our evaluation will ensure that the Panda gives the same pain scores as the traditional methods.

DETAILED DESCRIPTION:
The purpose of this study is to ensure that Panda, a smartphone-based pain assessment tool, can be used effectively by children after surgery and that the pain scores it obtains agree with the scores obtained using traditional methods of pain assessment. In particular the aim is to show agreement (a) between pain scores obtained using Panda and pain scores obtained using the Faces Pain Scale-Revised for 4-12 year olds and (b) between pain scores obtained using Panda and pain scores obtained using the Coloured Analogue Scale (CAS) for 5-18 year olds.

We will recruit children between 4 and 18 years old, in general good health, who are scheduled for surgery. We will exclude any child who has a psychiatric diagnosis, developmental delay or brain injury, significant visual impairment or psychomotor dysfunction.

This study is taking place in the Post-anesthetic Care Unit (PACU) at BC Children's Hospital. We will recruit 200 children in total. The study procedures include the following:

Stage 1 - pre-clinical usability study: we will conduct a series of participatory design sessions with nurses in the PACU and with 20 children in the Surgical Day Care Unit (SDCU)

Stage 2 - clinical validation study: children will be asked to rate their pain using both the Panda and a traditional tool (which is used first will be decided randomly); during this stage, children will also be asked their opinion (e.g. which tool they preferred using and about any problems they experienced using either tool).

All scores will be recorded on the Panda device and extracted at the end of each day. No pain medication will be administered on the basis of a pain score obtained using the Panda.

Panda will be compared with the traditional method (FPS-R and CAS) within 3 different age groups (4-8, 8-12 and 12-18), using the following criteria: practicality, based on failure rates in obtaining pain scores from Panda compared with traditional method; preference for Panda compared with traditional method; agreement between the Panda score and the traditional score.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a surgical procedure for which there is an anticipated post-surgical pain model
* Age 4 - 18 years
* ASA I-III, not requiring admission to PICU
* Written parental/guardian informed consent and subject informed assent when required (subject age ≥ 7 years)

Exclusion Criteria:

* Children who have not undergone a surgical procedure (e.g. MRI, X-ray or endoscopy patients)
* Inability or refusal to provide informed consent/assent
* Developmental delay, neurological injury or psychomotor dysfunction
* Children who have a significant visual impairment or have undergone eye surgery

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Concordance between the electronic and paper versions of the FPS-R and CAS pain scales | Up to 2 hours following surgery
  The study aims to measure concordance between the (a) pain scores obtained using Panda and pain scores obtained using the Faces Pain Scale-Revised for 4-12 year olds and (b) pain scores obtained using Panda and pain scores obtained using the Coloured Analogue Scale (CAS) for 5-18 year olds.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ansermino, Study Director — UBC/Medicine, Faculty of/Anesthesiology, Pharmacology & Therapeutics; Gillian Lauder, Principal Investigator — UBC/Medicine, Faculty of/Anesthesiology, Pharmacology & Therapeutics
Locations (1):
- British Columbia Children's Hospital Department of Anesthesia, Vancouver, British Columbia, Canada